CLINICAL TRIAL: NCT06480019
Title: IPT-based Group Intervention by Non-specialist for Improvement of Depressive Symptoms in Community Young Adults in Brazil: a Randomized Clinical Trial
Brief Title: IPT-based Group Intervention by Non-specialist for Improvement of Depressive Symptoms in Community Young Adults in Brazil
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Neusa Sica da Rocha, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0283
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Depression; Interpersonal Relations
MeSH Terms: conditions — Depression | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Participants that receive psychotherapy
  Interventions: Behavioral: Interpersonal psychotherapy
- Waiting list (No Intervention): Participants that are waiting for intervention

INTERVENTIONS:
Behavioral: Interpersonal psychotherapy — Interpersonal psychotherapy is a first-line treatment and can also be used for the prevention of depression.
  Arms: Intervention

SUMMARY:
Major depressive disorder is a highly prevalent, recurrent, and debilitating disease, the third cause of years of lost life in the world, and it may be the most common disease in 2030, according to the World Health Organization (WHO). Furthermore, it's also related to decreased quality of life and high mortality. Interpersonal psychotherapy (IPT) is a first-line treatment and can also be used for the prevention of depression.

This randomized controlled clinical trial is planned to have 50 participants randomized between an interventional and a control group (waiting list). Our study covers young adults (18 to 24 years old) with depression. Participants will be invited by social media to undergo treatment in an IPT group. The intervention group will be separated into groups with up to 10 participants, with a weekly meeting for eight weeks. The intervention will focus on interpersonal relationships within the model of IPT and will be held by a university student and a doctor trained in IPT.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (between 18 and 24 years old)
* Young adults who work, live or study in Porto Alegre
* PHQ ≥ 5 - without suicide ideation

Exclusion Criteria:

* Maniac or hypomanic episode
* Psychotic Syndrome
* Substance Abuse
* Suicide Risk or Ideation

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Pre-treatment, Week 1 to 8
  The Hospital Anxiety and Depression Scale consists of 14 items, of which 7 assess anxiety and 7 assess depression. Each item is scored from 0 to 3, and each subscale has a maximum score of 21 points with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | Pre-treatment, Week 1 to 8
  The PHQ-9 is a self-administered instrument that quantitatively assesses the severity of depressive symptoms over the past two weeks. It consists of nine items corresponding to the diagnostic criteria for major depressive disorder in the DSM-IV. Each item is scored on a 4-point Likert scale (0 = not at all to 3 = nearly every day), resulting in a score ranging from 0 to 27.
Social support scale (MOS-SSS) | Pre-treatment, Week 1 to 8
  The Medical Outcomes Study Social Support Survey (MOS-SSS) measures each individual's perceptions of personal support. The scale comprises five support factors (emotional, informational, material, affective, and positive social interaction). Higher scores indicate greater perceived support.
Quality of Life (WHOQOL-BREF) | Pre-treatment, Week 1 to 8
  The WHOQOL-BREF is a scale with 26 items that measure quality of life. It includes two general items and 24 items representing four domains (physical, psychological, social relationships, and environmental).
Clinical Global Impression (CGI) | Pre-treatment, Week 1 to 8
  The Clinical Global Impressions (CGI) scale is an instrument that enables clinicians to assess the overall severity of the illness, the change in clinical status over time, and the effectiveness of the intervention used. Its score can range from 1 (not ill) to 7 (extremely ill).
Beck Depression Inventory (BDI) | Pre-treatment; Week 1-8
  It's a self-report instrument and assesses the presence and severity of depressive symptoms. It consists of 21 items describing cognitive, affective, and somatic manifestations of depression. Each item is scored in a Likert scale ranging from 0 to 3, varying from 0 to 63 points

OTHER OUTCOMES:
Resilience (CD-RISC-10) | Pre-treatment, Week 1 to 8
  The 10-item Connor-Davidson Resilience Scale (CD-RISC-10) is an abbreviated version of the original 25-item scale. It measures the capacity to adapt physically, mentally, and spiritually to the circumstances imposed by life. The 10 items are scored from 0 to 4, yielding a total score from 0 to 40. Higher scores indicate higher levels of resilience.
Psychotherapy side effects (UE-ATR checklist) | Week 1 to 8
  It allows finding, classifying and discriminating between undesirable effects, adverse reactions to treatment and side effects of psychotherapy, based on the assessment of possible domains of unwanted effects in severity and relationship with the treatment.
Childhood Trauma Questionnaire (CTQ) | Week 1
  The Childhood Trauma Questionnaire is a retrospective self-report instrument designed to assess experiences of childhood abuse and neglect. It consists of 28 items scored on a 5-point Likert scale, measuring five domains of maltreatment: emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect.
Life Stressful Events Questionnaire | Week 1 to 8
  It assesses through closed questions, with dichotomous answers (yes vs. no), covering stressful life events.
Attachment (RSQ) | Week 1 and 8
  The Relationship Scales Questionnaire (RSQ) assesses attachment styles in interpersonal relationships. It consists of 30 items describing thoughts and feelings in close relationships. Respondents rate their agreement with each item on a 5-point Likert scale. It assesses attachment through 30 declarative statements that express feelings and thoughts related to close relationships with people.
Eysenck Personality Questionnaire-Revised (EPQR-A) | Pre-treatment; Week 1-8
  It is a self-administered questionnaire composed of 24 items divided into four domains: the three dimensions of personality (neuroticism, extraversion, and psychoticism) and a validity scale (social desirability).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital for Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil